CLINICAL TRIAL: NCT05969912
Title: Effects of Instrument Assisted Soft Tissue Mobilization and Bowen Technique in Chronic Low Back Pain of Fibromyalgia
Brief Title: Effects of Instrument Assisted Soft Tissue Mobilization and Bowen Technique in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01650 Anum Shaheen
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Fibromyalgia; Low Back Pain
Keywords: Bowen technique; Instrument assisted soft tissue mobilization
MeSH Terms: conditions — Fibromyalgia; Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston Technique (Instrumented assisted soft tissue mobilization) (Active Comparator): Graston technique + Conventional PT
  Interventions: Other: Graston Technique (Instrumented assisted soft tissue mobilization)
- Bowen's Technique (Soft tissue technique) (Active Comparator): Bowen's technique + Conventional PT
  Interventions: Other: Bowen's Technique(Soft tissue technique)

INTERVENTIONS:
Other: Graston Technique (Instrumented assisted soft tissue mobilization) — They would received Graston technique (Instrumented assisted soft tissue mobilization) as follow:
  Using lubricant (Vaseline) on the skin then a stainless steel instrument to relax the fascia and muscles. Frequency: 60 reps per min for 3 times/week for 3 consecutive weeks Intensity: moderate intensity (pain free) Time: 20 mins Type: Graston technique (Instrument assisted soft tissue mobilization)
  Additionally, the would receive Conventional PT :
  Ultrasound for 5 min Stretching exercises at lumbar : Frequency: 10 reps with 5 sec hold for 3 times/week for 3 weeks
  Arms: Graston Technique (Instrumented assisted soft tissue mobilization)
Other: Bowen's Technique(Soft tissue technique) — They would received Bowen's technique (Soft tissue technique) as follow:
  Bowen moves (15 - 20 times) with 2 mins gap between each set. Frequency: 3 times/week for 3 consecutive weeks Intensity: moderate intensity (pain free) Time: 20 mins Type: Bowen's technique (Soft tissue technique)
  Additionally, the would receive Conventional PT :
  Ultrasound for 5 min Stretching exercises at lumbar : Frequency: 10 reps with 5 sec hold for 3 times/week for 3 weeks
  Arms: Bowen's Technique (Soft tissue technique)

SUMMARY:
To compare the effects of Bowen's and Graston Technique in patients of chronic low back pain for reducing pain, enhancing lumbar range of motion and physical functioning and reducing depression.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic disease of idiopathic etiology, which is estimated to affect 2-4% of the population. It causes pain, stiffness, and tenderness in muscles, tendons, and joints, as well as sleep disturbances, fatigue, anxiety, depression, and alterations in intestinal functions. Chronic low back pain is a pain of more than 12 weeks limited to the lower area of the back .The chief complaint of a patient with fibromyalgia is widespread musculoskeletal pain which is bilateral and involves both upper and lower parts of the body. The pain may be localized initially, commonly in the neck and shoulders. The predominant description of the pain is muscle pain, but the patients may complain of joint pain as well .

Grastοn technique is an instrument assisted soft tissue treatment method (ІASTM) derived from the Cyriax1 cross-friction massage. Physіοtherapist strikes stainless steel instrument in a longitudinal dіrectіοn and in circular patterns at the treatment site. Many IASTM instruments including ASTYM, Fascial Abrasion Technique and Graston Technique etc. facilitates the healing process through increased fibroblast proliferation and increased collagen synthesis, maturation, and alignment.

Bowen Therapy is a dynamic fascial and muscle release approach, consisting of gentle cross-fiber movements applied to the fascia, muscles, tendons, muscle insertions, muscle septa, ligaments and viscera. It is named after Tom Bowen, who created a form of bodywork in Geelong, Australia and addresses the body as a whole unit rather than just the presenting symptoms.

The rationale for the use of these techniques is to identify the effects of IASTM and Bowen therapy in chronic low back pain of fibromyalgia and to analyze the additional effects of these techniques by reducing the hyperalgesia and excitability in central nervous system by working on the descending pain modulation system and to identify the most time effective treatment for chronic low back pain in fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 65 years
* Both Genders
* Patients with fibromyalgia were included in the study if they fulfilled criteria of the American college of rheumatology for fibromyalgia.
* Patients having chronic mechanical low back pain of more than three months

Exclusion Criteria:

* Patients with tumor, infection and major trauma to the spine causing fracture or disruption of spine.
* Patients with cauda equina syndrome
* Any neurological disorder
* Any previous spinal fusion surgery or spinal cord stimulation.
* Pregnant females

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Fibromyalgia impact questionnaire (FIQ) | 3 weeks
  The FIQ is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes. It has been designed to measure the components of health status that are believed to be most affected by FM.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 3 weeks
  The NPRS is a segmented numeric version of the visual analog scale which is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score.
Clinically useful depression outcome scale (CUDOS) | 3 weeks
  There are five categories in the empirically derived range of the depression severity of the CUDOS: scores of 11-20 represent minimal depression; 21-30, mild depression; 31-45, moderate depression; and 46 or higher, severe depression.
Bubble inclinometer | 3 weeks
  It is an instrument that measures the available range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- Daultala centre of CBR/CBID Daultala centre of CBR/CBID and (ALP Hospital Rawalpindi)., Gujar Khān, Pakistan

IPD SHARING:
Plan to Share IPD: No